CLINICAL TRIAL: NCT04028843
Title: SmartMoms in WIC: A Smartphone Intervention for WIC Mothers to Improve Nutrition and Weight Gain During Pregnancy
Brief Title: A Smartphone Intervention for WIC Mothers to Improve Nutrition and Weight Gain During Pregnancy
Acronym: SmartMomsinWIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Louisiana Department of Health (Unknown); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Leanne Redman, Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 2018-039; R01NR017644 (NIH)
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Weight Gain During Pregnancy

STUDY DESIGN:
Intervention Model Description: Parallel assigned stratified by maternal BMI and site
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WIC Nutrition (No Intervention): Participants will receive weight management advice and care through the standard Women, Infants, and Children program. They will also receive weekly health information related to pregnancy, birth, and infant health through a closed Facebook group.
- Healthy Beginnings (Experimental): Participants will receive the SmartMoms smartphone application, a wireless connected scale, and a Fitbit. The Healthy Beginnings program includes a 24 week intensive behavior modification program that targets healthy gestational weight gain through self-monitoring of weight and activity data, automated prescriptive feedback from the SmartMoms smartphone application, personalized feedback from counselors, and evidence-based behavioral intervention delivered throughout pregnancy.
  Interventions: Behavioral: Healthy Beginnings

INTERVENTIONS:
Behavioral: Healthy Beginnings — The program includes a 24 week intensive behavior modification program that targets healthy gestational weight gain through self-monitoring of weight and activity data, automated prescriptive feedback from the smartphone application, personalized feedback from counselors and, evidence-based behavioral intervention delivered throughout pregnancy.
  Arms: Healthy Beginnings

SUMMARY:
The study will test the effectiveness of a smartphone-based behavior modification program adapted for use in Women, Infants, and Children program in a state-wide, randomized controlled trial in 432 low-income women enrolled in the Louisiana Women, Infants, and Children program.

DETAILED DESCRIPTION:
The study is a multi-site randomized controlled trial, testing the effectiveness of the smartphone-based behavior modification program in pregnant women within the Louisiana Women, Infants, and Children program. Equal number of participants will be randomized to either the intervention or the control. Although the intervention itself lasts 24 weeks (only during pregnancy), women will be enrolled in this study for approximately 18 months, from the 10-16th week of pregnancy until 12 month postpartum follow-up. Study outcomes will be assessed at three visits during pregnancy (early, mid, and late,) and three visits postpartum (1, 6, and 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Less than 16 weeks gestational age at screening visit
* Have a BMI of 18.5 to 40 kg/m2
* Expecting a singleton pregnancy
* Certified to receive Women, Infants, and Children services during current pregnancy
* Has smartphone with internet access
* Willing to be identifiable to other study participants in this study program

Exclusion Criteria:

* Smoking
* Drug or alcohol use
* Non-pregnancy related illness
* Hypertension at screening visit
* Current mental health issue or eating disorder
* Inability to complete a behavioral run-in task
* Plans to move out of the state in the next 18 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 351 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2025-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Redman, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual data can be shared with appropriate material/data use agreements but there are no current plans.

REFERENCES:
- [Derived] Kracht CL, Falkenhain K, Flanagan EW, Altazan AD, Cabre HE, Kebbe M, Woolf EK, Beyl R, Hsia DS, Apolzan JW, Redman L. Effect of a Pragmatic eHealth Behavioral Gestational Weight Gain Intervention on Household Chaos in Pregnant People of Lower Socioeconomic Status: Randomized Controlled Trial. JMIR Ment Health. 2026 Jan 8;13:e74146. doi: 10.2196/74146. PMID 41505178
- [Derived] Cabre HE, Falkenhain K, Altazan AD, Flanagan EW, Kracht CL, Sparks JR, Kebbe M, Woolf EK, Hsia DS, Gilmore LA, Beyl R, Apolzan JW, Redman LM. Examining the Impact of a Codeveloped Multicomponent Mobile eHealth Lifestyle Intervention on Physical Activity and Its Association With Gestational Weight Gain in Underserved Women: A Statewide Randomized Controlled Trial. J Med Internet Res. 2025 Nov 11;27:e73962. doi: 10.2196/73962. PMID 41218199
- [Derived] Kebbe M, Falkenhain K, Beyl R, Altazan AD, Flanagan EW, Kracht CL, Cabre HE, Woolf EK, Hsia DS, Apolzan JW, Redman LM. An eHealth Intervention in Pregnancy on Maternal Body Composition and Subsequent Perinatal Outcomes: A Randomized Trial. Obesity (Silver Spring). 2025 Sep;33(9):1680-1693. doi: 10.1002/oby.24357. Epub 2025 Jul 24. PMID 40707419
- [Derived] Flanagan EW, Altazan AD, Comardelle NR, Gilmore LA, Apolzan JW, St Romain J, Hardee JC, Puyau RS, Mayet CL, Beyl RA, Barlow SA, Bounds SS, Olson KN, Kennedy BM, Hsia DS, Redman LM. The Design of a Randomized Clinical Trial to Evaluate a Pragmatic and Scalable eHealth Intervention for the Management of Gestational Weight Gain in Low-Income Women: Protocol for the SmartMoms in WIC Trial. JMIR Res Protoc. 2020 Sep 10;9(9):e18211. doi: 10.2196/18211. PMID 32909954

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WIC Nutrition | Healthy Beginnings
Started | 172 | 179
Completed | 135 | 137
Not Completed | 37 | 42
Not completed — Lost to Follow-up | 32 | 39
Not completed — Adverse Event | 1 | 0
Not completed — Non-viable Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WIC Nutrition | Healthy Beginnings | Total
Number analyzed (Participants) | 172 | 179 | 351
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (6) | 27 (6) | 27 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 179 | 351
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 13 | 10 | 23
  Non-Hispanic White | 54 | 55 | 109
  Non-Hispanic Black | 95 | 106 | 201
  Mixed or Other | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Women Who Have Appropriate Gestational Weight Gain
Description: Number of pregnant women who gain appropriate weight during pregnancy as recommended by the Institute of Medicine Gestational Weight Gain guidelines
Time Frame: Approximately 6 months (from 10-16 weeks gestation to 35-38 weeks gestation)
Population: 46 participants enrolled in WIC Nutrition were missing primary outcome measures and are not included in primary and secondary outcome analysis (23 missing follow up weights, 4 discontinued intervention, 19 lost to follow up). 40 participants enrolled in Healthy Beginnings were missing primary outcome measures and are not included in primary and secondary outcome analysis (21 missing follow up weights, 2 discontinued intervention, 17 lost to follow up).
Measure: Count of Participants; unit: Participants
Arm/Group | WIC Nutrition | Healthy Beginnings
Number analyzed (Participants) | 126 | 139
Participants | 21 | 24

2. Secondary Outcome: Total Gestational Weight Gain
Description: Measured weight from 10-16 weeks gestation to 35-38 weeks gestation
Time Frame: Approximately 6 months (from 10-16 weeks gestation to 35-38 weeks gestation)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | WIC Nutrition | Healthy Beginnings
Number analyzed (Participants) | 126 | 139
kilograms | 10.9 [9.9 to 11.9] | 9.5 [8.5 to 10.5]

3. Secondary Outcome: Gestational Weight Gain Per Week
Description: Weight measured from 10-16 weeks gestation to 35-38 weeks gestation divided by the number of weeks between measures.
Time Frame: Approximately 6 months (from 10-16 weeks gestation to 35-38 weeks gestation)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | WIC Nutrition | Healthy Beginnings
Number analyzed (Participants) | 126 | 139
kilograms | 0.53 [0.48 to 0.57] | 0.46 [0.42 to 0.50]

ADVERSE EVENTS:
Time Frame: Approximately 18 months (from 10-16th week of pregnancy until 12 month postpartum follow up)
Arm/Group | WIC Nutrition | Healthy Beginnings
All-Cause Mortality (participants affected / at risk) | 0/172 | 0/179
Serious Adverse Events (participants affected / at risk) | 36/172 | 26/179
Other Adverse Events (participants affected / at risk) | 110/172 | 134/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WIC Nutrition (N=172) | Healthy Beginnings (N=179)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Benign tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder puncture (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal Bleeding (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2)
Blunt abdominal trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COVID-19 (General disorders) | 1 (1) | 0 (0)
Dehydration (Vascular disorders) | 1 (1) | 1 (1)
Ear infection (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Elevated heart rate (Cardiac disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Gallbladder infection (Infections and infestations) | 1 (1) | 0 (0)
Gallstones (Gastrointestinal disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Incompetent cervix (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Leg lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Low fetal activity (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Steroid allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 7 (7)
Preterm contractions (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 2 (2)
Preterm delivery (Pregnancy, puerperium and perinatal conditions) | 12 (12) | 6 (6)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WIC Nutrition (N=172) | Healthy Beginnings (N=179)
Anemia (Blood and lymphatic system disorders) | 11 (11) | 24 (24)
COVID-19 (General disorders) | 14 (14) | 18 (18)
Depression (Psychiatric disorders) | 12 (12) | 16 (16)
Gestational diabetes (Endocrine disorders) | 13 (13) | 13 (13)
Headache (Nervous system disorders) | 20 (22) | 18 (20)
Heartburn (Gastrointestinal disorders) | 17 (17) | 26 (26)
Hypertension (Vascular disorders) | 15 (16) | 20 (23)
Low iron (Blood and lymphatic system disorders) | 10 (11) | 14 (14)
Nausea/vomiting (Gastrointestinal disorders) | 52 (54) | 69 (74)
Urinary tract infection (Renal and urinary disorders) | 9 (9) | 9 (10)
Vaginal delivery pain (Pregnancy, puerperium and perinatal conditions) | 12 (12) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT04028843/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT04028843/SAP_001.pdf